CLINICAL TRIAL: NCT01404780
Title: Comparison of the Glidescope and Macintosh Laryngoscope for Double Lumen Endotracheal Tube Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-0270-B
Record Dates: First submitted 2011-06-21; First posted 2011-07-28 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Lung Disease
Keywords: Double lumen ET intubation; Laryngoscope; Lung Surgery
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The GlideScope (GVL) (Experimental)
  Interventions: Device: GlideScope (GVL)
- Macintosh direct laryngoscope (MDL) (Active Comparator)
  Interventions: Device: Macintosh Direct Laryngoscope (MDL)

INTERVENTIONS:
Device: GlideScope (GVL) — The Glidescope (GVL) has not been extensively studied for double lumen tube intubation. The GVL may be particularly useful for patients with difficult airways as it has a camera attached to the blade.
  Arms: The GlideScope (GVL)
Device: Macintosh Direct Laryngoscope (MDL) — Current standard of care at UHN for 50 years
  Arms: Macintosh direct laryngoscope (MDL)

SUMMARY:
Patients undergoing chest surgery often require insertion of a breathing tube (double lumen tube) after they are unconscious. The double lumen tube enables the anaesthetist to ventilate (assist breathing) one lung at a time. The other lung is partially deflated to enable enough space for the surgeon to perform the procedure. The breathing tube is inserted with a laryngoscope (blade with a light at the end) so the vocal cords can be seen. This is standard medical practise. Two laryngoscopes are commonly used at Toronto General Hospital to insert the tube. The Macintosh laryngoscope has been is use for over 50 years and the Glidescope for over 10 years. Both devices have been extensively researched for single lumen tubes insertion and found to be very safe and effective. Research is limited to say which of the two laryngoscope is the most effective for double lumen tubes.

DETAILED DESCRIPTION:
The Glidescope (GVL) has been extensively studied for single lumen tube intubation and found to be a very safe and useful device. It is a particularly useful for patients with difficult airways as it has a camera attached to the blade. Despite being used for double lumen tube (DLT) intubations, research of its effectiveness and safety, is lacking. The study aims to determine the speed and safety of the GVL for DLT insertion. This information will assist anaesthetists in choosing the appropriate laryngoscope for DLT intubation of their patients.

ELIGIBILITY:
Inclusion Criteria:

Population: planned elective lung surgery requiring general anaesthesia with a double lumen endotracheal intubation, signed informed patient consent.

Exclusion Criteria:

* Previous failed intubation,
* history of difficult intubation or anticipated difficult intubation (2 risk factors of mallampati score 3 or greater,
* incisor gap < 3.5cm, thyromental distance < 6.5cm,
* reduced neck extension and flexion),
* alternative method of intubation indicated eg rapid sequence intubation,
* fibreoptic intubation,
* contra-indication to a left double lumen tube eg endobronchial tumor,
* significant deviation or compression of the trachea and bronchi.,
* contraindication to one lung ventilation eg severe hypoxia or pulmonary hypertension,
* anticipated difficult bag mask ventilation,
* symptomatic gastro-oesophageal reflux,
* oral/pharyngeal/laryngeal carcinoma,
* loose teeth,
* allergy to rocuronium, BMI > 40.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Time to intubation (laryngoscope or DLT inserted between patient's lips to DLT placement in the trachea and laryngoscope withdrawal) | Number of minutes (0-2) that is required to intubate will be recorded, if a 2nd attempt is required, duration to successfull intubation will be recorded in minutes.
  Patients will be randomized to either MDL or GVL. If the first attempt fails to intubate within 2 minutes the anesthetist will remove the laryngoscope and provide mask ventilation. The second intubation attempt the anesthetist is encouraged to use the same randomized laryngoscope however, if the treating anesthetist feels a different device and technique will have a higher success rate they can perform that technique on the second attempt regardless of the randomized device. Anesthetists will complete a questionnaire after intubation.

SECONDARY OUTCOMES:
Time to lung isolation, difficulty of the procedure, complication to the patients | From the beginning of the operative procedure through to 24 hours postoperatively
  Information about the procedure (times and complications) will be collected and documented by the study Anesthetist and questionnaires completed at the end of the 24hr postoperative period. Visits: patients will be followed up for a 24 hour period either on ward or by telephone if discharged, and assessed for sore throat, hoarseness, trauma to mouth and lips, dental damage and swallowing difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Van Rensburg, MD, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada